CLINICAL TRIAL: NCT02576613
Title: Modified Psychodynamic Psychotherapy for Patients With Schizophrenia - a Randomized Controlled Trial
Brief Title: Modified Psychodynamic Psychotherapy for Patients With Schizophrenia
Acronym: MPP-S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: International Psychoanalytic University Berlin (Other)
Responsible Party: Principal Investigator, Christiane Montag MD, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EA1/200/15
Record Dates: First submitted 2015-10-08; First posted 2015-10-15 (Estimated); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MPP-S (Experimental): at least 30 weekly sessions of modified psychodynamic psychotherapy
  Interventions: Other: MPP-S
- standard therapy (TAU) (Experimental): clinical standard treatment, including supportive therapeutic contacts, pharmacotherapy, creative and occupational therapies, psychoeducation, group therapies, excluding structured individual or group psychotherapy
  Interventions: Other: TAU

INTERVENTIONS:
Other: MPP-S — > 30 weekly sessions of modified psychodynamic psychotherapy in addition to standard treatment
  Other Names: Modified psychodynamic psychotherapy
  Arms: MPP-S
Other: TAU — standard medical treatment without structured psychotherapeutic intervention
  Other Names: treatment as usual
  Arms: standard therapy (TAU)

SUMMARY:
A randomized controlled, prospective, two-armed, mono-centric, assessor-blinded clinical trial will serve to generate preliminary data on the efficacy and safety of modified psychodynamic therapy (MPP-S) in stabilized patients after the first or subsequent episodes of schizophrenia or schizoaffective disorder.

DETAILED DESCRIPTION:
Rationale: Compared to the existing evidence for other psychotherapy methods like cognitive-behavioral psychotherapy or family interventions, the scientific basis of psychodynamic psychotherapy for psychoses is weak with respect to randomized-controlled research. Its encouragement by expert opinion and the broad application of this method stands in sharp contrast to the apparent lack of research interest regarding its efficacy and safety and the fact that more people suffering from schizophrenic spectrum disorders will hopefully embark on psychotherapy in the coming years.

The aim of the presented study is therefore on the one hand to explore the efficacy and safety of modified psychodynamic psychotherapy (MPP-S) in a randomized controlled study design. On the other hand, psychodynamic assumptions regarding the treatment of psychotic persons shall be elucidated in an explorative part of the study. For this purpose, a newly developed manual of modified psychodynamic psychotherapy for psychoses will be inaugurated.

Primary objective of the study is to determine whether the administration of MPP-S in addition to standard treatment (=treatment as usual: TAU) will lead to an improvement of psychosocial functioning in outpatients with schizophrenia and schizo-affective disorder compared to standard treatment.

Secondary objectives refer to the question, whether symptom domains and necessity of hospital treatment, as well as interpersonal functioning and subjective recovery might be impacted by MPP-S compared to TAU alone. Moreover, theoretical assumptions about possible psychodynamic mechanisms of action of MPP-S led to exploratory hypotheses, which are to be tested.

Safety and tolerability of the psychodynamic intervention will be evaluated by acquisition of safety data during study visits, but also by continuous monitoring of participants' condition after every treatment session and clinical contact.

Additional exploratory objectives of this study deal with the question, whether cerebral functional activity and connectivity within the so-called "Default-Mode-Network" (DMN) measured with fMRI are influenced by psychodynamic psychotherapy in the intervention group compared to the control condition. Moreover, changes of functional correlates of social cognition before and after psychotherapy or TAU will be compared between groups using a video-based social-cognitive task during fMRI.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizo-affective disorder according to DSM-IV-TR
* Age 18-64 years
* Sufficient German language competence
* Written informed consent
* Consent to audio recording of psychotherapy sessions and video-taping of assessment interviews at study visits

Exclusion Criteria:

* Organic brain disorder
* Relevant somatic disorder impairing cerebral function
* Relevant abuse alcohol and illegal drugs as assessed by a current or previous indication for treatment for addiction
* Inability to understand and comply with the requirements of the study and to give written informed consent
* CDSS-item for suicidal ideation is marked >/= 2
* Massive agitation or current endangerment of others

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2015-10; Primary Completion 2021-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
psychosocial functioning | 6 months
  Primary endpoint is the Mini-ICF-APP (=Mini-International Classification of Functioning for limitations of Activities and Participation in Psychological disorders) as a measure of disorders of capacity as defined by the International Classification of Functioning
psychosocial functioning | 12 months
  Primary endpoint is the Mini-ICF-APP (=Mini-International Classification of Functioning for limitations of Activities and Participation in Psychological disorders) as a measure of disorders of capacity as defined by the International Classification of Functioning
psychosocial functioning | 24 months
  Primary endpoint is the Mini-ICF-APP (=Mini-International Classification of Functioning for limitations of Activities and Participation in Psychological disorders) as a measure of disorders of capacity as defined by the International Classification of Functioning
psychosocial functioning | 36 months
  Primary endpoint is the Mini-ICF-APP (=Mini-International Classification of Functioning for limitations of Activities and Participation in Psychological disorders)

SECONDARY OUTCOMES:
psychotic symptom severity | 6 months
  psychotic symptoms measured by Positive and Negative Syndrome Scale (PANSS)
psychotic symptom severity | 12 months
  psychotic symptoms measured by Positive and Negative Syndrome Scale (PANSS)
psychotic symptom severity | 24 months
  psychotic symptoms measured by Positive and Negative Syndrome Scale (PANSS)
psychotic symptom severity | 36 months
  psychotic symptoms measured by Positive and Negative Syndrome Scale (PANSS)
depressive symptom severity | 6 months
  depressive symptoms measured by Calgary Depression Scale for Schizophrenia
depressive symptom severity | 12 months
  depressive symptoms measured by Calgary Depression Scale for Schizophrenia
depressive symptom severity | 24 months
  depressive symptoms measured by Calgary Depression Scale for Schizophrenia
depressive symptom severity | 36 months
  depressive symptoms measured by Calgary Depression Scale for Schizophrenia
necessity of hospital treatment | 6 months
  necessity of hospital (inpatient) treatment, measured cumulative days in hospital per year
necessity of hospital treatment | 12 months
  necessity of hospital (inpatient) treatment, measured cumulative days in hospital per year
necessity of hospital treatment | 24 months
  necessity of hospital (inpatient) treatment, measured cumulative days in hospital per year
necessity of hospital treatment | 36 months
  necessity of hospital (inpatient) treatment, measured cumulative days in hospital per year
general symptom severity | 6 months
  Clinical Global Impression (CGI Severity und Improvement)
general symptom severity | 12 months
  Clinical Global Impression (CGI Severity und Improvement)
general symptom severity | 24 months
  Clinical Global Impression (CGI Severity und Improvement)
general symptom severity | 36 months
  Clinical Global Impression (CGI Severity und Improvement)
psychic "structure" | 6 months
  Axes II-VI (relationships, conflicts, structure) of the Operationalized Psychodynamic Diagnostics (OPD)
psychic "structure" | 12 months
  Axes II-VI (relationships, conflicts, structure) of the Operationalized Psychodynamic Diagnostics (OPD)
psychic "structure" | 24 months
  Axes II-VI (relationships, conflicts, structure) of the Operationalized Psychodynamic Diagnostics (OPD)
psychic "structure" | 36 months
  Axes II-VI (relationships, conflicts, structure) of the Operationalized Psychodynamic Diagnostics (OPD)
metacognitive function | 6 months
  Metacognition Assessment Scale-Abbreviated (MAS-A)
metacognitive function | 12 months
  Metacognition Assessment Scale-Abbreviated (MAS-A)
metacognitive function | 24 months
  Metacognition Assessment Scale-Abbreviated (MAS-A)
metacognitive function | 36 months
  Metacognition Assessment Scale-Abbreviated (MAS-A)
cognitive and emotional mentalization | baseline
  Movie for the Assessment of Social Cognition (MASC)
cognitive and emotional mentalization | 12 months
  Movie for the Assessment of Social Cognition (MASC)
"mentalized affectivity" and emotional awareness | 6 months
  Levels of Emotional Awareness Scale (LEAS)
"mentalized affectivity" and emotional awareness | 12 months
  Levels of Emotional Awareness Scale (LEAS)
"mentalized affectivity" and emotional awareness | 24 months
  Levels of Emotional Awareness Scale (LEAS)
self-rated ability to solve interpersonal problems | 6 months
  Inventory of Interpersonal Problems (IIP-D)
self-rated ability to solve interpersonal problems | 12 months
  Inventory of Interpersonal Problems (IIP-D)
self-rated ability to solve interpersonal problems | 24 months
  Inventory of Interpersonal Problems (IIP-D)
self-rated ability to solve interpersonal problems | 36 months
  Inventory of Interpersonal Problems (IIP-D)
ability to make subjective sense of psychotic experiences | 6 months
  Questionnaire to assess subjective meaning in psychosis (SuSi)
ability to make subjective sense of psychotic experiences | 12 months
  Questionnaire to assess subjective meaning in psychosis (SuSi)
ability to make subjective sense of psychotic experiences | 24 months
  Questionnaire to assess subjective meaning in psychosis (SuSi)
ability to make subjective sense of psychotic experiences | 36 months
  Questionnaire to assess subjective meaning in psychosis (SuSi)
Changes in cerebral functional activity, connectivity, structure of social cognitive and default-mode networks from Baseline | baseline
  BOLD-contrast, structure
Changes in cerebral functional activity, connectivity, structure of social cognitive and default-mode networks from Baseline | 24 months
  BOLD-contrast, structure

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Montag, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Psychiatrische Universitätsklinik der Charité im St. Hedwig Krankenhaus, Berlin, Germany